CLINICAL TRIAL: NCT03926143
Title: An Open-label, Multicenter Rollover Study to Provide Continued Treatment With Anetumab Ravtansine for Participants With Solid Tumors Who Were Enrolled in Previous Bayer-sponsored Studies
Brief Title: A Clinical Study of Anetumab Ravtansine in Adults With Solid Tumors Who Have Been Treated in Previous Bayer-sponsored Anetumab Ravtansine Studies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to strategic company decisions, the development of anetumab ravtansine was stopped.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20322; 2019-000061-20 (EudraCT Number)
Record Dates: First submitted 2019-04-23; First posted 2019-04-24 (Actual); Results first posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Solid Tumors
Keywords: Solid tumors; Mesothelin; Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — anetumab ravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cancer patients (Experimental): Adult patients with solid cancer who received anetumab-ravtansine treatment in a completed Bayer study
  Interventions: Drug: BAY94-9343 (Anetumab ravtansine)

INTERVENTIONS:
Drug: BAY94-9343 (Anetumab ravtansine) — BAY94-9343 (Anetumab ravtansine) will be administered as specified in the parent studies
  Other Names: Anti-mesothelin antibody, Maytansinoid tubulin inhibitor DM4

SUMMARY:
The purpose of this study is to enable patients with solid tumors, who received anetumab ravtansine in a Bayer-sponsored clinical trial, to continue treatment after their respective study has been closed. The patients will be observed to collect information on how safe and efficient the drug is.

DETAILED DESCRIPTION:
The primary objective of the study is to collect long-term safety information on anetumab ravtansine and to enable patients, who received an anetumab ravtansine-containing treatment in any Bayer-sponsored anetumab ravtansine parent study, to continue the treatment. The secondary objective is to further investigate the efficacy of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Participants ongoing in an applicable Bayer-sponsored anetumab ravtansine parent study at the time of its planned study closure.
* For on-treatment participants: participant is eligible to receive the next dose of study intervention per the parent study protocol.
* For on-treatment participants: any ongoing adverse events that require temporary treatment interruption must be resolved to baseline grade or assessed as stable and not requiring further treatment interruption. For applicable studies: should treatment be permanently interrupted in the parent study, participants may be enrolled in the follow-up portion of the rollover study.

Exclusion Criteria:

* For on-treatment participants: a positive serum pregnancy test.
* For on-treatment participants: use of one or more of the prohibited medications listed in the respective parent study protocol.
* Participants who are receiving standard-of-care agent(s) but not anetumab ravtansine in the parent study, and are able to receive standard-of-care agent outside of the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - University of Chicago, Chicago, Illinois
  - National Cancer Institute - Maryland, Bethesda, Maryland
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Mary Crowley Medical Research Center, Dallas, Texas
- Hôpital de la Timone - Marseille, Marseille, France
- ASST Grande Ospedale Metropolitano Niguarda, Milan, Lombardy, Italy
- Samodzielny Publiczny Wojewodzki Szpital Zespolony, Szczecin-Zdunowo, Poland

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 7 study centers in 4 countries worldwide between 03-Jun-2019 (first participant first visit) and 18-May-2022 (last participant last visit). Entering participants had to have been treated with anetumab ravtansine in an applicable Bayer sponsored anetumab ravtansine parent study.
Pre-assignment Details: A total of 10 participants were screened in this study; of whom 9 participants started study treatment and 1 participant was a screening failure.
Groups:
- Anetumab Ravtansine: Adult participants with solid tumors who received anetumab-ravtansine treatment as monotherapy, or in combination with gemcitabine in an applicable Bayer-sponsored anetumab ravtansine study.
  8 participants received anetumab ravtansine monotherapy and 1 participant received anetumab ravtansine in combination with gemcitabine. Pooled results were reported.
Period: Overall Study
Arm/Group | Anetumab Ravtansine
Started | 9
Completed | 0
Not Completed | 9
Not completed — Physician Decision | 3
Not completed — Subject decision: Covid-19 Pandemic related | 1
Not completed — Adverse Event | 2
Not completed — Progressive disease | 3

BASELINE CHARACTERISTICS:
Arm/Group | Anetumab Ravtansine
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (16.2) [lower limit 16.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Ethnicity [Count of Participants; unit: Participants]
  Unknown or Not Reported | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With TEAEs, TESAEs and Drug-related TEAEs and TESAEs
Description: Treatment emergent adverse events (TEAEs) were defined as AEs starting or worsening during the treatment period. The treatment period extended from the first date of study treatment in this study until the safety follow-up (30 days after the last administration of study treatment). TESAEs: Treatment emergent serious adverse events.
Time Frame: Approximately 3 years (from first study treatment until safety follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | Anetumab Ravtansine
Number analyzed (Participants) | 9
Participants
  Any TEAE | 9
  Serious TEAE | 2
  Any study drug-related TEAE | 8
  Any study drug-related Serious TEAE | 0

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) defined as the time from first treatment in this study until death from any cause. Data on survival were collected by the site. Time frame was reduced due to early termination of the study. Table reports Kaplan-Meier median with Brookmeyer-Crowley confidence intervals. Number (%) of participants with event: 5 (55.6%) and Number (%) of participants censored: 4 (44.4%).
Time Frame: Approximately 3 years (from first study treatment until safety follow-up)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Anetumab Ravtansine
Number analyzed (Participants) | 9
Months
  25th percentile | 17.6 [6.9 to 34.1]
  Median | 34.1 [6.9 to NA] — "Not applicable" indicates value cannot be estimated due to censored data.
  75th percentile | NA [28.5 to NA] — "Not applicable" indicates value cannot be estimated due to censored data.

ADVERSE EVENTS:
Time Frame: For TEAE: After the first study intervention up to 30 days after the end of study intervention, approximately 3 years. For the all-cause mortality: considering all deaths that occurred at any time during the study before the last contact, up to approximately 3 years.
Description: Per the Statistical Analysis Plan, pooled ("by overall") results were reported and no differentiation on treatment of anetumab-ravtansine as monotherapy or in combination with gemcitabine.
Arm/Group | Anetumab Ravtansine
All-Cause Mortality (participants affected / at risk) | 5/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anetumab Ravtansine (N=9)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (2)
Oedema peripheral (General disorders) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anetumab Ravtansine (N=9)
Anaemia (Blood and lymphatic system disorders) | 5 (10)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3)
Pericardial effusion (Cardiac disorders) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Corneal disorder (Eye disorders) | 1 (1)
Corneal epithelial microcysts (Eye disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 2 (3)
Conjunctivitis (Infections and infestations) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Amylase increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 1 (3)
Blood bilirubin increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (2)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 2 (3)
Neutrophil count decreased (Investigations) | 1 (2)
Weight decreased (Investigations) | 1 (4)
Transaminases increased (Investigations) | 1 (1)
Schirmer's test abnormal (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 2 (6)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (6)
Gynaecomastia (Reproductive system and breast disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the small sample size and heterogeneous population, survival distributions and the extent of long-term survival in the applicable populations cannot be reliably estimated from the study results.

Overall results were reported. Pooling was done because there is only a single patient treated with combination and no summary tables on a single patient.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/43/NCT03926143/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT03926143/SAP_001.pdf